CLINICAL TRIAL: NCT05975671
Title: Reducing Empiric VAncomycin Use in Pediatric Suspected Sepsis (REVAMP-Sepsis)
Brief Title: Reducing Empiric VAncomycin Use in Pediatric Suspected Sepsis
Acronym: REVAMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Healthcare of Atlanta (Other); St. Louis Children's Hospital (Other); Johns Hopkins University (Other); University of Pennsylvania (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-019410; U54CK000610-02-00 (Other Grant/Funding Number: Centers for Disease Control); U54CK000610 (NIH)
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Sepsis; Sepsis Mrsa; Sepsis Bacteremia; Antimicrobial - Induced Nephropathy; Sepsis, Severe; Septic Shock; Septic Syndrome
Keywords: Sepsis; Vancomycin use; methicillin-resistant Staphylococcus aureus (MRSA); Antibiotic Stewardship; Implementation science
MeSH Terms: conditions — Sepsis; Shock, Septic; Toxemia

STUDY DESIGN:
Intervention Model Description: Multicenter, mixed methods, implementation science study with a quasi-experimental design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICU Clinicians and Sepsis stakeholders (Other): Clinicians and sepsis stakeholders in the participating sites will be primarily recruited via email. During the course of this multifaceted intervention:
  * All the PICU (Pediatric Intensive Care Unit) prescribing clinicians and sepsis stakeholders in the participating sites will receive clinical guidelines, unit-level feedback reports, and education on Vancomycin use during the intervention.
  * Investigators will perform semi-structured interviews with 90 PICU clinicians and sepsis stakeholders.
  * Surveys will be sent to all eligible clinicians, estimated to be up to 2500 individuals across the 4 sites. These structured surveys will be done at baseline and at 9 months post-implementation.
  Interventions: Behavioral: Multifaceted de-implementation strategy to reduce vancomycin overuse
- PICU Patients with suspected sepsis (No Intervention): Research procedures involving patients will be limited to medical record review. This medical record review will help inform the intervention directed at PICU clinicians/stakeholders and the assessment of study outcomes. Approximately 50,000 patients will participate in the study. Data elements will be collected at each site and stored as password-protected Comma-separated values (CSV) files. These files will not contain any direct Protected Health Information (PHI) but will contain elements of date (e.g., date of admission, date of suspected sepsis episode). The study Identification (ID) number will be used to identify each unique patient. Each site will collect and store data in compliance with the Children's Hospital of Philadelphia (CHOP) and local Institutional Review Board (IRB) policies.

INTERVENTIONS:
Behavioral: Multifaceted de-implementation strategy to reduce vancomycin overuse — * Clinical guidelines and group-level feedback on vancomycin use will be provided to clinicians/sepsis stakeholders at each site.
  * The semi-structured interviews will be performed by a trained member of the research team, under the supervision of a medical sociologist who is one of the co-investigators. A semi-structured interview guide will be used during the interviews. Interviews will be recorded and transcribed, then uploaded to a qualitative analysis software for management and coding. Names will not be recorded, and pseudonyms will be used in notes, communications about the study, and any presentations. Verbal consent will be obtained before conducting and recording the interviews.
  * The surveys will be performed using REDCap survey software, and participation will be voluntary. No identifiers will be collected.
  Other Names: Mixed methods intervention
  Arms: PICU Clinicians and Sepsis stakeholders

SUMMARY:
The goal of this quasi-experimental interventional study is to determine the effectiveness of a multifaceted stewardship intervention in reducing overall vancomycin use in five tertiary care Pediatric Intensive Care Units (PICU).

There are two groups of subjects in this study: PICU clinicians/sepsis stakeholders and patients admitted to one of the participating PICUs during the study period. The intervention will at a minimum include:

* Implementation of a clinical guideline indicating when vancomycin should and should not be used
* Unit-level feedback on overall vancomycin use within and across centers
* Clinician education.

DETAILED DESCRIPTION:
Vancomycin is among the most commonly prescribed antibiotics in United States children's hospitals, and inappropriate use of vancomycin is common. Given the high prevalence of acute kidney injury associated with vancomycin of up to 25%, reducing vancomycin overuse is a key opportunity to reduce preventable patient harm.

The primary objective of this study is to determine the effectiveness of a multifaceted stewardship intervention in reducing overall vancomycin use in five tertiary care PICUs. This intervention will be informed by baseline data surrounding vancomycin use and infections due to organisms requiring vancomycin therapy which will allow selective use of vancomycin, as well as a concurrent mixed methods process and formative evaluation to inform implementation of the intervention.

During the baseline period, Electronic Health Record (EHR) data will be used to retrospectively quantify unit-level vancomycin use over 24 months (measured as vancomycin days of therapy [DOT]/1000 patient days), as well as the frequency of vancomycin use and prevalence of infections due to organisms requiring vancomycin therapy among patients with suspected and confirmed sepsis.

During the post-intervention period, which will last approximately 24 months, a multifaceted stewardship intervention to reduce vancomycin use informed by these baseline data, including:

* The creation of a consensus guideline for vancomycin use;
* Ad hoc education related to vancomycin overuse, and;
* Unit-level feedback on vancomycin prescribing. The feedback on vancomycin use will be provided to clinicians at each site, both within their site (to compare to past performance) and across sites (to compare local performance to the performance of other sites).

This intervention will be locally adapted by the investigative team and sepsis stakeholders at each site. Data from the EHR will be used to assess vancomycin use (DOT/1000 patient days), as well as the secondary outcomes. Investigators will perform semi-structured interviews and repeat surveys 9 months after the implementation of the intervention. This mixed-methods process and formative evaluation will help investigators understand which elements of implementation were successful and which were not.

ELIGIBILITY:
Patient Inclusion Criteria:

* Admitted to one of the participating PICUs during the study period

Patient Exclusion Criteria:

* None

Clinician Inclusion Criteria:

1. PICU prescribing clinician (including attending physicians, fellows, residents, nurse practitioners, and physician assistants) OR sepsis stakeholder (leader of sepsis quality improvement work, medical director) at one of the participating sites at the time the survey is deployed
2. Age ≥ 18 years old
3. Employed by one of the participating sites

Clinician Exclusion Criteria:

1. Volunteers or other non-employee hospital staff
2. Limited English proficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52500 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in vancomycin use | Baseline to 5 years
  Vancomycin use will be measured as DOT per 1000 PICU patient days, measured monthly. Every day in which one or more doses of parenteral vancomycin is administered is classified as one vancomycin DOT. Every day or portion of a day a patient is admitted to the PICU is classified as one PICU patient day.

SECONDARY OUTCOMES:
Change in rate of suspected and confirmed sepsis episodes per 1000 PICU patient days. | Baseline to 5 years
  Change in the rate of suspected and confirmed sepsis episodes in which new or persistent respiratory, renal, cardiovascular, or hematologic organ dysfunction occur at day 3 and at day 7.
PICU all-cause mortality | Up to 3 years
  All-cause mortality will be measured at 30 days following sepsis onset as a proportion of suspected and confirmed sepsis episodes. Only one episode of suspected or confirmed sepsis will be counted in this measure.
PICU length of stay | Up to 3 years
  Time elapsed between a patient's admission into the PICU and discharge from the PICU.
Hospital length of stay | Up to 3 years
  Time elapsed between a patient's hospital admittance and discharge.
30-day PICU readmission | Within 30 days of discharge from a PICU admission
  Readmission to the PICU is defined as an admission to the PICU occurring within 30 days following discharge from an admission in which there was one or more episodes of suspected or confirmed sepsis. Only one episode of suspected or confirmed sepsis will be counted in this measure. Patients without a readmission to the index hospital or health system will be counted as no readmission, due to the inability to assess readmissions to outside institutions.
30-day hospital readmission | Within 30 days of discharge from a hospital admission
  The percentage of patients that are readmitted to the hospital within 30 days following discharge from an admission in which there was one or more episodes of suspected or confirmed sepsis. Only one episode of suspected or confirmed sepsis will be counted in this measure.
Use of other broad-spectrum antibiotics | Up to 5 years
  Cefepime, ceftriaxone, and piperacillin-tazobactam DOT/1000 PICU days, measured monthly (as a non-equivalent dependent variable).
Use of other anti-MRSA antibiotics | Up to 5 years
  Linezolid, Ceftaroline, clindamycin, and trimethoprim-sulfamethoxazole in DOT/1000 patient days, measured monthly (as a balancing measure to evaluate any increase in other anti-MRSA antibiotics that may occur as an unintended consequence of reducing vancomycin use).
Prevalence of infections due to organisms requiring vancomycin | Up to 5 years
  Microbiologic outcome measures will focus on the prevalence of vancomycin-requiring organisms in the suspected and confirmed sepsis cohorts, and will also be measured relative to the frequency of empiric vancomycin administration and compliance with the guideline.

OTHER OUTCOMES:
Adoption of intervention | Onset of intervention to 2 years
  Adoption, the decision to adhere to the guideline for vancomycin use, will be measured as the proportion of sepsis episodes in which the clinician adhered to the guideline based on medical record review. Adoption will be evaluated in a 10% random sample of sepsis episodes each month by chart review.
Appropriateness of intervention | Onset of intervention to 2 years
  Appropriateness, the perceived compatibility of the intervention to the PICU practice setting, will be measured during surveys and semi-structured interviews using the Likert Scale; where 1 = completely disagree and 5 = completely agree.
Acceptability of intervention | Onset of intervention to 2 years
  Acceptability, how well the intervention was received by the PICU clinicians will be measured during surveys and semi-structured interviews using the Likert Scale; where 1 = completely disagree and 5 = completely agree.
Measure of feasibility of intervention | Onset of intervention to 2 years
  Feasibility, the extent to which the intervention can be carried out in the setting, will be determined in collaboration with our local stakeholders but may include the proportion of PICU clinicians who attend educational sessions and/or unit-based meetings during which vancomycin use data is reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Chiotos, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (4):
- United States (4):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
This study was initiated prior to the NIH Data Management and Sharing Policy update that was released on January 25, 2023.

REFERENCES:
- [Background] Kissoon N, Reinhart K, Daniels R, Machado MFR, Schachter RD, Finfer S. Sepsis in Children: Global Implications of the World Health Assembly Resolution on Sepsis. Pediatr Crit Care Med. 2017 Dec;18(12):e625-e627. doi: 10.1097/PCC.0000000000001340. PMID 28914721
- [Background] Weiss SL, Peters MJ, Alhazzani W, Agus MSD, Flori HR, Inwald DP, Nadel S, Schlapbach LJ, Tasker RC, Argent AC, Brierley J, Carcillo J, Carrol ED, Carroll CL, Cheifetz IM, Choong K, Cies JJ, Cruz AT, De Luca D, Deep A, Faust SN, De Oliveira CF, Hall MW, Ishimine P, Javouhey E, Joosten KFM, Joshi P, Karam O, Kneyber MCJ, Lemson J, MacLaren G, Mehta NM, Moller MH, Newth CJL, Nguyen TC, Nishisaki A, Nunnally ME, Parker MM, Paul RM, Randolph AG, Ranjit S, Romer LH, Scott HF, Tume LN, Verger JT, Williams EA, Wolf J, Wong HR, Zimmerman JJ, Kissoon N, Tissieres P. Surviving Sepsis Campaign International Guidelines for the Management of Septic Shock and Sepsis-Associated Organ Dysfunction in Children. Pediatr Crit Care Med. 2020 Feb;21(2):e52-e106. doi: 10.1097/PCC.0000000000002198. PMID 32032273
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Crit Care Med. 2017 Mar;45(3):486-552. doi: 10.1097/CCM.0000000000002255. PMID 28098591
- [Background] Tamma PD, Avdic E, Li DX, Dzintars K, Cosgrove SE. Association of Adverse Events With Antibiotic Use in Hospitalized Patients. JAMA Intern Med. 2017 Sep 1;177(9):1308-1315. doi: 10.1001/jamainternmed.2017.1938. PMID 28604925
- [Background] Same RG, Hsu AJ, Cosgrove SE, Klein EY, Amoah J, Hersh AL, Kronman MP, Tamma PD. Antibiotic-Associated Adverse Events in Hospitalized Children. J Pediatric Infect Dis Soc. 2021 May 28;10(5):622-628. doi: 10.1093/jpids/piaa173. PMID 33452808
- [Background] Hensgens MP, Goorhuis A, Dekkers OM, Kuijper EJ. Time interval of increased risk for Clostridium difficile infection after exposure to antibiotics. J Antimicrob Chemother. 2012 Mar;67(3):742-8. doi: 10.1093/jac/dkr508. Epub 2011 Dec 6. PMID 22146873
- [Background] Bell BG, Schellevis F, Stobberingh E, Goossens H, Pringle M. A systematic review and meta-analysis of the effects of antibiotic consumption on antibiotic resistance. BMC Infect Dis. 2014 Jan 9;14:13. doi: 10.1186/1471-2334-14-13. PMID 24405683
- [Background] Lovegrove MC, Geller AI, Fleming-Dutra KE, Shehab N, Sapiano MRP, Budnitz DS. US Emergency Department Visits for Adverse Drug Events From Antibiotics in Children, 2011-2015. J Pediatric Infect Dis Soc. 2019 Nov 6;8(5):384-391. doi: 10.1093/jpids/piy066. PMID 30137509
- [Background] Downes KJ, Cowden C, Laskin BL, Huang YS, Gong W, Bryan M, Fisher BT, Goldstein SL, Zaoutis TE. Association of Acute Kidney Injury With Concomitant Vancomycin and Piperacillin/Tazobactam Treatment Among Hospitalized Children. JAMA Pediatr. 2017 Dec 4;171(12):e173219. doi: 10.1001/jamapediatrics.2017.3219. Epub 2017 Dec 4. PMID 28973124
- [Background] Navalkele B, Pogue JM, Karino S, Nishan B, Salim M, Solanki S, Pervaiz A, Tashtoush N, Shaikh H, Koppula S, Koons J, Hussain T, Perry W, Evans R, Martin ET, Mynatt RP, Murray KP, Rybak MJ, Kaye KS. Risk of Acute Kidney Injury in Patients on Concomitant Vancomycin and Piperacillin-Tazobactam Compared to Those on Vancomycin and Cefepime. Clin Infect Dis. 2017 Jan 15;64(2):116-123. doi: 10.1093/cid/ciw709. Epub 2016 Oct 20. PMID 27986669
- [Background] Rutter WC, Cox JN, Martin CA, Burgess DR, Burgess DS. Nephrotoxicity during Vancomycin Therapy in Combination with Piperacillin-Tazobactam or Cefepime. Antimicrob Agents Chemother. 2017 Jan 24;61(2):e02089-16. doi: 10.1128/AAC.02089-16. Print 2017 Feb. PMID 27895019
- [Background] Dethlefsen L, Huse S, Sogin ML, Relman DA. The pervasive effects of an antibiotic on the human gut microbiota, as revealed by deep 16S rRNA sequencing. PLoS Biol. 2008 Nov 18;6(11):e280. doi: 10.1371/journal.pbio.0060280. PMID 19018661
- [Background] McKamy S, Hernandez E, Jahng M, Moriwaki T, Deveikis A, Le J. Incidence and risk factors influencing the development of vancomycin nephrotoxicity in children. J Pediatr. 2011 Mar;158(3):422-6. doi: 10.1016/j.jpeds.2010.08.019. PMID 20888013
- [Background] Sinclair EA, Yenokyan G, McMunn A, Fadrowski JJ, Milstone AM, Lee CK. Factors associated with acute kidney injury in children receiving vancomycin. Ann Pharmacother. 2014 Dec;48(12):1555-62. doi: 10.1177/1060028014549185. Epub 2014 Sep 3. PMID 25186624
- [Background] Ragab AR, Al-Mazroua MK, Al-Harony MA. Incidence and predisposing factors of vancomycin-induced nephrotoxicity in children. Infect Dis Ther. 2013 Jun;2(1):37-46. doi: 10.1007/s40121-013-0004-8. Epub 2013 Mar 26. PMID 25135822
- [Background] Fiorito TM, Luther MK, Dennehy PH, LaPlante KL, Matson KL. Nephrotoxicity With Vancomycin in the Pediatric Population: A Systematic Review and Meta-Analysis. Pediatr Infect Dis J. 2018 Jul;37(7):654-661. doi: 10.1097/INF.0000000000001882. PMID 29280786
- [Background] Feiten HDS, Okumura LM, Martinbiancho JK, Andreolio C, da Rocha TS, Antonacci Carvalho PR, Pedro Piva J. Vancomycin-associated Nephrotoxicity and Risk Factors in Critically Ill Children Without Preexisting Renal Injury. Pediatr Infect Dis J. 2019 Sep;38(9):934-938. doi: 10.1097/INF.0000000000002391. PMID 31232892
- [Background] Bradley JS, Byington CL, Shah SS, Alverson B, Carter ER, Harrison C, Kaplan SL, Mace SE, McCracken GH Jr, Moore MR, St Peter SD, Stockwell JA, Swanson JT; Pediatric Infectious Diseases Society and the Infectious Diseases Society of America. The management of community-acquired pneumonia in infants and children older than 3 months of age: clinical practice guidelines by the Pediatric Infectious Diseases Society and the Infectious Diseases Society of America. Clin Infect Dis. 2011 Oct;53(7):e25-76. doi: 10.1093/cid/cir531. Epub 2011 Aug 31. PMID 21880587
- [Background] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710
- [Background] Tribble AC, Lee BR, Flett KB, Handy LK, Gerber JS, Hersh AL, Kronman MP, Terrill CM, Sharland M, Newland JG; Sharing Antimicrobial Reports for Pediatric Stewardship (SHARPS) Collaborative. Appropriateness of Antibiotic Prescribing in United States Children's Hospitals: A National Point Prevalence Survey. Clin Infect Dis. 2020 Nov 5;71(8):e226-e234. doi: 10.1093/cid/ciaa036. PMID 31942952
- [Background] Brogan TV, Thurm C, Hersh AL, Gerber JS, Smith MJ, Shah SS, Courter JD, Patel SJ, Parker SK, Kronman MP, Lee BR, Newland JG. Variability in Antibiotic Use Across PICUs. Pediatr Crit Care Med. 2018 Jun;19(6):519-527. doi: 10.1097/PCC.0000000000001535. PMID 29533352
- [Background] Blinova E, Lau E, Bitnun A, Cox P, Schwartz S, Atenafu E, Yau Y, Streitenberger L, Parshuram CS, Marshall J, Seto W. Point prevalence survey of antimicrobial utilization in the cardiac and pediatric critical care unit. Pediatr Crit Care Med. 2013 Jul;14(6):e280-8. doi: 10.1097/PCC.0b013e31828a846d. PMID 23823209
- [Background] Williams MC, Obermeier H, Hurst AL, Saporta-Keating SR, Pearce K, MacBrayne CE, Child J, Parker SK. Hospital-wide Description of Clinical Indications for Pediatric Anti-infective Use. Clin Ther. 2019 Aug;41(8):1605-1611.e0. doi: 10.1016/j.clinthera.2019.05.008. Epub 2019 Jun 11. PMID 31196642
- [Background] Mermel LA. Respiratory protection for healthcare workers caring for COVID-19 patients. Infect Control Hosp Epidemiol. 2020 Sep;41(9):1064-1065. doi: 10.1017/ice.2020.175. Epub 2020 Apr 23. No abstract available. PMID 32321614
- [Background] Metlay JP, Waterer GW, Long AC, Anzueto A, Brozek J, Crothers K, Cooley LA, Dean NC, Fine MJ, Flanders SA, Griffin MR, Metersky ML, Musher DM, Restrepo MI, Whitney CG. Diagnosis and Treatment of Adults with Community-acquired Pneumonia. An Official Clinical Practice Guideline of the American Thoracic Society and Infectious Diseases Society of America. Am J Respir Crit Care Med. 2019 Oct 1;200(7):e45-e67. doi: 10.1164/rccm.201908-1581ST. PMID 31573350
- [Background] Levine DP. Vancomycin: a history. Clin Infect Dis. 2006 Jan 1;42 Suppl 1:S5-12. doi: 10.1086/491709. PMID 16323120
- [Background] Weiner-Lastinger LM, Abner S, Benin AL, Edwards JR, Kallen AJ, Karlsson M, Magill SS, Pollock D, See I, Soe MM, Walters MS, Dudeck MA. Antimicrobial-resistant pathogens associated with pediatric healthcare-associated infections: Summary of data reported to the National Healthcare Safety Network, 2015-2017. Infect Control Hosp Epidemiol. 2020 Jan;41(1):19-30. doi: 10.1017/ice.2019.297. Epub 2019 Nov 25. PMID 31762428
- [Background] Waters CD, Caraccio J. Rate of positive cultures necessitating definitive treatment in patients receiving empiric vancomycin therapy. Infect Control Hosp Epidemiol. 2018 Aug;39(8):989-990. doi: 10.1017/ice.2018.123. Epub 2018 Jun 12. PMID 29893660
- [Background] Jones M, Jernigan JA, Evans ME, Roselle GA, Hatfield KM, Samore MH. Vital Signs: Trends in Staphylococcus aureus Infections in Veterans Affairs Medical Centers - United States, 2005-2017. MMWR Morb Mortal Wkly Rep. 2019 Mar 8;68(9):220-224. doi: 10.15585/mmwr.mm6809e2. PMID 30845116
- [Background] Jones BE, Jones MM, Huttner B, Stoddard G, Brown KA, Stevens VW, Greene T, Sauer B, Madaras-Kelly K, Rubin M, Goetz MB, Samore M. Trends in Antibiotic Use and Nosocomial Pathogens in Hospitalized Veterans With Pneumonia at 128 Medical Centers, 2006-2010. Clin Infect Dis. 2015 Nov 1;61(9):1403-10. doi: 10.1093/cid/civ629. Epub 2015 Jul 29. PMID 26223995
- [Background] Jones BE, Brown KA, Jones MM, Huttner BD, Greene T, Sauer BC, Madaras-Kelly K, Rubin MA, Bidwell Goetz M, Samore MH. Variation in Empiric Coverage Versus Detection of Methicillin-Resistant Staphylococcus aureus and Pseudomonas aeruginosa in Hospitalizations for Community-Onset Pneumonia Across 128 US Veterans Affairs Medical Centers. Infect Control Hosp Epidemiol. 2017 Aug;38(8):937-944. doi: 10.1017/ice.2017.98. Epub 2017 Jun 21. PMID 28633678
- [Background] Sutter DE, Milburn E, Chukwuma U, Dzialowy N, Maranich AM, Hospenthal DR. Changing Susceptibility of Staphylococcus aureus in a US Pediatric Population. Pediatrics. 2016 Apr;137(4):e20153099. doi: 10.1542/peds.2015-3099. Epub 2016 Mar 1. PMID 26933211
- [Background] Kim NH, Koo HL, Choe PG, Cheon S, Kim M, Lee MJ, Jung Y, Park WB, Song KH, Kim ES, Bang JH, Kim HB, Park SW, Kim NJ, Oh MD, Kim EC. Inappropriate continued empirical vancomycin use in a hospital with a high prevalence of methicillin-resistant Staphylococcus aureus. Antimicrob Agents Chemother. 2015 Feb;59(2):811-7. doi: 10.1128/AAC.04523-14. Epub 2014 Nov 17. PMID 25403664
- [Background] Davies P, Evans C, Kanthimathinathan HK, Lillie J, Brierley J, Waters G, Johnson M, Griffiths B, du Pre P, Mohammad Z, Deep A, Playfor S, Singh D, Inwald D, Jardine M, Ross O, Shetty N, Worrall M, Sinha R, Koul A, Whittaker E, Vyas H, Scholefield BR, Ramnarayan P. Intensive care admissions of children with paediatric inflammatory multisystem syndrome temporally associated with SARS-CoV-2 (PIMS-TS) in the UK: a multicentre observational study. Lancet Child Adolesc Health. 2020 Sep;4(9):669-677. doi: 10.1016/S2352-4642(20)30215-7. Epub 2020 Jul 9. PMID 32653054
- [Background] Choe PG, Koo HL, Yoon D, Bae JY, Lee E, Hwang JH, Song KH, Park WB, Bang JH, Kim ES, Kim HB, Park SW, Oh MD, Kim NJ. Effect of an intervention targeting inappropriate continued empirical parenteral vancomycin use: a quasi-experimental study in a region of high MRSA prevalence. BMC Infect Dis. 2018 Apr 16;18(1):178. doi: 10.1186/s12879-018-3081-1. PMID 29661158
- [Background] Junior MS, Correa L, Marra AR, Camargo LF, Pereira CA. Analysis of vancomycin use and associated risk factors in a university teaching hospital: a prospective cohort study. BMC Infect Dis. 2007 Aug 1;7:88. doi: 10.1186/1471-2334-7-88. PMID 17678541
- [Background] Rhee C, Kadri SS, Dekker JP, Danner RL, Chen HC, Fram D, Zhang F, Wang R, Klompas M; CDC Prevention Epicenters Program. Prevalence of Antibiotic-Resistant Pathogens in Culture-Proven Sepsis and Outcomes Associated With Inadequate and Broad-Spectrum Empiric Antibiotic Use. JAMA Netw Open. 2020 Apr 1;3(4):e202899. doi: 10.1001/jamanetworkopen.2020.2899. PMID 32297949
- [Background] Jones BE, Ying J, Stevens V, Haroldsen C, He T, Nevers M, Christensen MA, Nelson RE, Stoddard GJ, Sauer BC, Yarbrough PM, Jones MM, Goetz MB, Greene T, Samore MH. Empirical Anti-MRSA vs Standard Antibiotic Therapy and Risk of 30-Day Mortality in Patients Hospitalized for Pneumonia. JAMA Intern Med. 2020 Apr 1;180(4):552-560. doi: 10.1001/jamainternmed.2019.7495. PMID 32065604
- [Background] Hranjec T, Rosenberger LH, Swenson B, Metzger R, Flohr TR, Politano AD, Riccio LM, Popovsky KA, Sawyer RG. Aggressive versus conservative initiation of antimicrobial treatment in critically ill surgical patients with suspected intensive-care-unit-acquired infection: a quasi-experimental, before and after observational cohort study. Lancet Infect Dis. 2012 Oct;12(10):774-80. doi: 10.1016/S1473-3099(12)70151-2. Epub 2012 Aug 28. PMID 22951600
- [Background] Hoelen DW, Tjan DH, van Vugt R, van der Meer YG, van Zanten AR. Severe local vancomycin induced skin necrosis. Br J Clin Pharmacol. 2007 Oct;64(4):553-4. doi: 10.1111/j.1365-2125.2007.02897.x. Epub 2007 Apr 10. No abstract available. PMID 17425624
- [Background] Fridkin SK, Edwards JR, Courval JM, Hill H, Tenover FC, Lawton R, Gaynes RP, McGowan JE Jr; Intensive Care Antimicrobial Resistance Epidemiology (ICARE) Project and the National Nosocomial Infections Surveillance (NNIS) System Hospitals. The effect of vancomycin and third-generation cephalosporins on prevalence of vancomycin-resistant enterococci in 126 U.S. adult intensive care units. Ann Intern Med. 2001 Aug 7;135(3):175-83. doi: 10.7326/0003-4819-135-3-200108070-00009. PMID 11487484
- [Background] Brownlee S, Chalkidou K, Doust J, Elshaug AG, Glasziou P, Heath I, Nagpal S, Saini V, Srivastava D, Chalmers K, Korenstein D. Evidence for overuse of medical services around the world. Lancet. 2017 Jul 8;390(10090):156-168. doi: 10.1016/S0140-6736(16)32585-5. Epub 2017 Jan 9. PMID 28077234
- [Background] Norton WE, Chambers DA, Kramer BS. Conceptualizing De-Implementation in Cancer Care Delivery. J Clin Oncol. 2019 Jan 10;37(2):93-96. doi: 10.1200/JCO.18.00589. Epub 2018 Nov 8. No abstract available. PMID 30407894
- [Background] Niven DJ, Mrklas KJ, Holodinsky JK, Straus SE, Hemmelgarn BR, Jeffs LP, Stelfox HT. Towards understanding the de-adoption of low-value clinical practices: a scoping review. BMC Med. 2015 Oct 6;13:255. doi: 10.1186/s12916-015-0488-z. PMID 26444862
- [Background] Barlam TF, Childs E, Zieminski SA, Meshesha TM, Jones KE, Butler JM, Damschroder LJ, Goetz MB, Madaras-Kelly K, Reardon CM, Samore MH, Shen J, Stenehjem E, Zhang Y, Drainoni ML. Perspectives of Physician and Pharmacist Stewards on Successful Antibiotic Stewardship Program Implementation: A Qualitative Study. Open Forum Infect Dis. 2020 Jun 15;7(7):ofaa229. doi: 10.1093/ofid/ofaa229. eCollection 2020 Jul. PMID 32704510
- [Background] Newland JG, Stach LM, De Lurgio SA, Hedican E, Yu D, Herigon JC, Prasad PA, Jackson MA, Myers AL, Zaoutis TE. Impact of a Prospective-Audit-With-Feedback Antimicrobial Stewardship Program at a Children's Hospital. J Pediatric Infect Dis Soc. 2012 Sep;1(3):179-86. doi: 10.1093/jpids/pis054. Epub 2012 Jul 12. PMID 26619405
- [Background] Aizawa Y, Suwa J, Higuchi H, Fukuoka K, Furuichi M, Kaneko T, Morikawa Y, Okazaki K, Shimizu N, Horikoshi Y. Antimicrobial Stewardship Program in a Pediatric Intensive Care Unit. J Pediatric Infect Dis Soc. 2018 Aug 17;7(3):e156-e159. doi: 10.1093/jpids/piy031. PMID 29688433
- [Background] Cantey JB, Wozniak PS, Pruszynski JE, Sanchez PJ. Reducing unnecessary antibiotic use in the neonatal intensive care unit (SCOUT): a prospective interrupted time-series study. Lancet Infect Dis. 2016 Oct;16(10):1178-1184. doi: 10.1016/S1473-3099(16)30205-5. Epub 2016 Jul 22. PMID 27452782
- [Background] Woods-Hill CZ, Fackler J, Nelson McMillan K, Ascenzi J, Martinez DA, Toerper MF, Voskertchian A, Colantuoni E, Klaus SA, Levin S, Milstone AM. Association of a Clinical Practice Guideline With Blood Culture Use in Critically Ill Children. JAMA Pediatr. 2017 Feb 1;171(2):157-164. doi: 10.1001/jamapediatrics.2016.3153. PMID 27942705
- [Background] Prusaczyk B, Swindle T, Curran G. Defining and conceptualizing outcomes for de-implementation: key distinctions from implementation outcomes. Implement Sci Commun. 2020 Apr 30;1:43. doi: 10.1186/s43058-020-00035-3. eCollection 2020. PMID 32885200
- [Background] Davey P, Marwick CA, Scott CL, Charani E, McNeil K, Brown E, Gould IM, Ramsay CR, Michie S. Interventions to improve antibiotic prescribing practices for hospital inpatients. Cochrane Database Syst Rev. 2017 Feb 9;2(2):CD003543. doi: 10.1002/14651858.CD003543.pub4. PMID 28178770
- [Background] Lorencatto F, Charani E, Sevdalis N, Tarrant C, Davey P. Driving sustainable change in antimicrobial prescribing practice: how can social and behavioural sciences help? J Antimicrob Chemother. 2018 Oct 1;73(10):2613-2624. doi: 10.1093/jac/dky222. PMID 30020464
- [Background] Pandolfo AM, Horne R, Jani Y, Reader TW, Bidad N, Brealey D, Enne VI, Livermore DM, Gant V, Brett SJ; INHALE WP2 Study Group. Understanding decisions about antibiotic prescribing in ICU: an application of the Necessity Concerns Framework. BMJ Qual Saf. 2022 Mar;31(3):199-210. doi: 10.1136/bmjqs-2020-012479. Epub 2021 Jun 7. PMID 34099497
- [Background] Wunderink RG, Srinivasan A, Barie PS, Chastre J, Dela Cruz CS, Douglas IS, Ecklund M, Evans SE, Evans SR, Gerlach AT, Hicks LA, Howell M, Hutchinson ML, Hyzy RC, Kane-Gill SL, Lease ED, Metersky ML, Munro N, Niederman MS, Restrepo MI, Sessler CN, Simpson SQ, Swoboda SM, Guillamet CV, Waterer GW, Weiss CH. Antibiotic Stewardship in the Intensive Care Unit. An Official American Thoracic Society Workshop Report in Collaboration with the AACN, CHEST, CDC, and SCCM. Ann Am Thorac Soc. 2020 May;17(5):531-540. doi: 10.1513/AnnalsATS.202003-188ST. PMID 32356696
- [Background] Cressman AM, MacFadden DR, Verma AA, Razak F, Daneman N. Empiric Antibiotic Treatment Thresholds for Serious Bacterial Infections: A Scenario-based Survey Study. Clin Infect Dis. 2019 Aug 30;69(6):930-937. doi: 10.1093/cid/ciy1031. PMID 30535310
- [Background] Szymczak JE, Muller BM, Shakamuri NS, Hamilton KW, Gerber JS, Laguio-Vila M, Dumyati GK, Fridkin SK, Guh AY, Reddy SC, Lautenbach E; CDC Prevention Epicenters Program. Prescriber perceptions of fluoroquinolones, extended-spectrum cephalosporins, and Clostridioides difficile infection. Infect Control Hosp Epidemiol. 2020 Aug;41(8):914-920. doi: 10.1017/ice.2020.183. Epub 2020 May 29. PMID 32468967
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426